CLINICAL TRIAL: NCT04553107
Title: Reducing Healthcare Costs in Older Adults by Deprescribing Unnecessary, Harmful, and Costly Medications
Brief Title: Reducing Costs by Deprescribing Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Blue Cross Blue Shield (Other)
Responsible Party: Principal Investigator, Holly M Holmes, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2019-410
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Polypharmacy; Deprescribing; Adverse Drug Reaction
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deprescribing Intervention (Experimental)
  Interventions: Behavioral: Deprescribing Intervention
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Deprescribing Intervention — An individualized deprescribing intervention will be created by a pharmacist working with a patient to identify harmful, costly, and unnecessary medications to be reduced. The intervention will include a plan and monitoring for up to 3 months to reduce medication use.
  Arms: Deprescribing Intervention
Behavioral: Usual Care — The usual care arm will receive the current standard of care, which includes medication reconciliation by a clinic nurse at the time of their appointment. Nurses review all medications and answer medication-related questions, and refer medication questions to the healthcare provider for further discussion when necessary.
  Arms: Usual Care

SUMMARY:
The purpose of the study is to implement a pharmacist-led deprescribing intervention for adults 65 and older taking 10 or more medications at University of Texas (UT) Physicians clinics and to assess the effect of the pharmacist intervention on the incidence of adverse drug reactions, emergency room visits, and hospitalizations as well as costs to the patient and to the healthcare system in adults 65 and older taking 10 or more medications treated at UT Physicians.

ELIGIBILITY:
Inclusion Criteria:

- taking 10 or more regular medications

Exclusion Criteria:

* not receiving primary care at UT Physicians

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 419 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Adverse Drug Reactions (ADR) | 3 months post enrollment
  Patient-reported side effects and adverse events potentially attributable to medication, rated for the likelihood of ADR by an independent reviewer based on the Naranjo algorithm.
Adverse Drug Reactions | 6 months post enrollment
  Patient-reported side effects and adverse events potentially attributable to medication, rated for the likelihood of ADR by an independent reviewer based on the Naranjo algorithm.
Adverse Drug Reactions | 12 months post enrollment
  Patient-reported side effects and adverse events potentially attributable to medication, rated for the likelihood of ADR by an independent reviewer based on the Naranjo algorithm.
Healthcare Cost | 3 months post enrollment
  Healthcare cost based on utilization of clinic visits, emergency room visits, and hospitalizations, based on patient report with specific costs obtained when possible from the Health Information Exchange.
Healthcare Cost | 6 months post enrollment
  Healthcare cost based on utilization of clinic visits, emergency room visits, and hospitalizations, based on patient report with specific costs obtained when possible from the Health Information Exchange.
Healthcare Cost | 12 months post enrollment
  Healthcare cost based on utilization of clinic visits, emergency room visits, and hospitalizations, based on patient report with specific costs obtained when possible from the Health Information Exchange.

SECONDARY OUTCOMES:
Medication use | At enrollment
  Number and name of each medication a participant is taking.
Medication cost | 3 months post enrollment
  Average wholesale price of each medication taken by a participant, determined using reference software.
Medication cost | 6 months post enrollment
  Average wholesale price of each medication taken by a participant, determined using reference software.
Medication cost | 12 months post enrollment
  Average wholesale price of each medication taken by a participant, determined using reference software.
QOL | Baseline
  Quality of life as measured by the EQ5D scale.This scale is numbered from 0 to 100. 100 means the best health you can imagine. 0 means the worst health you can imagine.
QOL | 12 months post enrollment
  Quality of life as measured by the EQ5D scale.This scale is numbered from 0 to 100. 100 means the best health you can imagine. 0 means the worst health you can imagine.

CONTACTS AND LOCATIONS:
Overall Officials: Holly M Holmes, MD,MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States